CLINICAL TRIAL: NCT00684203
Title: Phase II Study of SCH 530348 in Subjects With Acute Coronary Syndrome
Brief Title: Trial to Assess the Safety and Effects of Vorapaxar in Japanese Subjects With Acute Coronary Syndrome (P04772; MK-5348-016)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P04772
Record Dates: First submitted 2008-05-22; First posted 2008-05-26 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-03

CONDITIONS: Atherosclerosis; Myocardial Ischemia; Myocardial Infarction
MeSH Terms: conditions — Atherosclerosis; Myocardial Ischemia; Myocardial Infarction | interventions — vorapaxar; Aspirin; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Vorapaxar 20 mg/1 mg (Experimental): Vorapaxar 20 mg loading dose + daily 1 mg maintenance dose + standard of care (Aspirin + Ticlopidine)
  Interventions: Drug: Vorapaxar; Drug: Aspirin; Drug: Clopidogrel
- Vorapaxar 20 mg/2.5 mg (Experimental): Vorapaxar 20 mg loading dose + daily 2.5 mg maintenance dose + standard of care (Aspirin + Ticlopidine)
  Interventions: Drug: Vorapaxar; Drug: Aspirin; Drug: Clopidogrel
- Vorapaxar 40 mg/1 mg (Experimental): Vorapaxar 40 mg loading dose + daily 1 mg maintenance dose + standard of care (Aspirin + Ticlopidine)
  Interventions: Drug: Vorapaxar; Drug: Aspirin; Drug: Clopidogrel
- Vorapaxar 40 mg/2.5 mg (Experimental): Vorapaxar 40 mg loading dose + daily 2.5 mg maintenance dose + standard of care (Aspirin + Ticlopidine)
  Interventions: Drug: Vorapaxar; Drug: Aspirin; Drug: Clopidogrel
- Placebo (Placebo Comparator): Placebo loading dose + daily placebo maintenance dose + standard of care (Aspirin + Ticlopidine)
  Interventions: Drug: Placebo; Drug: Aspirin; Drug: Clopidogrel

INTERVENTIONS:
Drug: Vorapaxar — Oral tablets; single 20-mg or 40-mg loading dose on first day followed by daily 1-mg or 2.5-mg maintenance dose for 59 days
  Arms: Vorapaxar 20 mg/1 mg; Vorapaxar 20 mg/2.5 mg; Vorapaxar 40 mg/1 mg; Vorapaxar 40 mg/2.5 mg
Drug: Placebo — Oral tablets; matching placebo for SCH 530348 loading and maintenance doses for 59 days
  Arms: Placebo
Drug: Aspirin — Loading dose of 75-325 mg on Day 1, then 75-100 mg once daily for 60 days.
  Other Names: ASA, acetylsalicylic acid
Drug: Clopidogrel — 100 mg two or three times daily for 60 days.

SUMMARY:
The study is designed to assess safety and effects of vorapaxar, when added to standard of care (aspirin and clopidigrel), in Japanese subjects with acute coronary syndrome. The study may also provide information about the effect of vorapaxar on preventing heart attack and stroke in this subject population.

DETAILED DESCRIPTION:
The study drug (loading dose) is administered at least 1 hour before catheterization for diagnostic imaging or percutaneous coronary interventions (PCI). The incidence of bleeding is thought to be an important index to assess the safety of this drug, therefore thrombolysis in myocardial infarction (TIMI) is evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 years or more with history of cardiac ischemia related chest discomfort of > 10 minutes duration < 24 hours prior to randomization, and having at least 1 of the following A or B. Participants who are planned to undergo PCI will be the target participants.

  * A: Positive biomarkers [Elevated troponin I or creatinine kinase MB isozyme greater than the site's upper limit of normal (ULN)] at or before registration
  * B: Electrocardiogram (ECG) changes: ST segment depression >= 0.1 mV (>=1 mm), or transient (<30 minutes) ST segment elevation >= 0.1 mV (>=1 mm) in at least 2 contiguous leads
* Willing to give appropriate informed consent and complete all study-related procedures, and able to adhere to dosing and all visit schedules.
* Women of child-bearing potential (all postmenarchal women who are <1 years menopausal or who have not had surgical sterilization or a hysterectomy are considered to be women of child-bearing potential) must agree to use a medically accepted method of contraception while receiving protocol-specified medication, and for 60 days after stopping the medication.

Exclusion Criteria:

* Pregnant and nursing mothers (premenopausal women should have a negative pregnancy test result confirmed before enrollment)
* Any serious illness or any condition that the investigator feels would pose a significant hazard to the participant if investigational therapy were initiated
* known hypersensitivity to any component of the current investigational product;
* Participation in a study of experimental therapy or use of any investigational drug within 30 days before enrollment
* Member of the staff personnel directly involved with this study;
* Family member of the investigational study staff;
* History of a bleeding diathesis, or evidence of active abnormal bleeding within 30 days before enrollment
* History of a hemorrhagic stroke at any time
* Severe hypertension (systolic blood pressure >200 mm Hg or diastolic blood pressure >110 mm Hg) while receiving therapy;
* Major surgery within 2 weeks prior to enrollment
* Known platelet count <100,000/mm^3
* Uncontrolled cardiac arrhythmia;
* Known impairment of renal function (serum creatinine >2.0 mg/dL [>176.8 umol/L]), dysproteinemia, nephrotic syndrome, or other renal disease;
* Active or chronic hepatobiliary or hepatic disease, or aspartate aminotransferase (AST) or alanine aminotransferase (ALT) activity more than two times greater than the upper limit of the laboratory reference range
* Anticipated staged PCI
* Concurrent or anticipated treatment with warfarin, factor Xa inhibitor, direct thrombin inhibitor, or antiplatelet agents except aspirin and ticlopidine after enrollment
* Anticipated intracoronary brachytherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2006-12-01 (Actual); Primary Completion 2007-10-01 (Actual); Study Completion 2007-10-01 (Actual)

REFERENCES:
- [Result] Goto S, Yamaguchi T, Ikeda Y, Kato K, Yamaguchi H, Jensen P. Safety and exploratory efficacy of the novel thrombin receptor (PAR-1) antagonist SCH530348 for non-ST-segment elevation acute coronary syndrome. J Atheroscler Thromb. 2010 Feb 26;17(2):156-64. doi: 10.5551/jat.3038. Epub 2010 Feb 3. PMID 20124733
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=P04772&kw=P04772&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 120 participants enrolled and randomized to treatment, 117 participants were treated with study drug. 92 participants underwent percutaneous coronary intervention (PCI) and 25 did not.
Groups:
- Vorapaxar 20 mg (PCI): Vorapaxar 20 mg as loading dose is administered to PCI participants as the initial dose. From Day 2, 1 mg or 2.5 mg once daily is administered as the maintenance dose for 59 days (total duration of 60 days).
- Vorapaxar 40 mg (PCI): Vorapaxar 40 mg as loading dose is administered to PCI participants as the initial dose. From Day 2, 1 mg or 2.5 mg once daily is administered as the maintenance dose for 59 days (total duration of 60 days).
- Placebo/Placebo (PCI): Placebo as loading dose is administered as the initial dose to PCI participants. From Day 2, placebo once daily is administered as the maintenance dose for 59 days (total duration of 60 days).
- Vorapaxar 20 mg (Non-PCI): Vorapaxar 20 mg as a loading dose is administered to non-PCI participants as the initial dose. From Day 2, 1 mg or 2.5 mg once daily is administered as the maintenance dose for 59 days (total duration 60 days).
- Vorapaxar 40 mg (Non-PCI): Vorapaxar 40 mg as loading dose is administered to non-PCI participants as the initial dose. From Day 2, 1 mg or 2.5 mg once daily is administered as the maintenance dose for 59 days (total duration of 60 days).
- Placebo/Placebo (Non-PCI): Placebo as loading dose is administered as the initial dose to non-PCI participants. From Day 2, placebo once daily is administered as the maintenance dose for 59 days (total duration of 60 days).
Period: Overall Study
Arm/Group | Vorapaxar 20 mg (PCI) | Vorapaxar 40 mg (PCI) | Placebo/Placebo (PCI) | Vorapaxar 20 mg (Non-PCI) | Vorapaxar 40 mg (Non-PCI) | Placebo/Placebo (Non-PCI)
Started | 40 | 31 | 21 | 6 | 17 | 2
Completed | 31 | 23 | 12 | 6 | 17 | 2
Not Completed | 9 | 8 | 9 | 0 | 0 | 0
Not completed — Adverse Event | 6 | 4 | 8 | 0 | 0 | 0
Not completed — Protocol-defined clinical event | 3 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 1 | 0 | 0 | 0
Not completed — Did not meet protocol eligibility | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vorapaxar 20 mg (PCI) | Vorapaxar 40 mg (PCI) | Placebo/Placebo (PCI) | Vorapaxar 20 mg (Non-PCI) | Vorapaxar 40 mg (Non-PCI) | Placebo/Placebo (Non-PCI) | Total
Number analyzed (Participants) | 40 | 31 | 21 | 6 | 17 | 2 | 117
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.3 (9.2) | 64.5 (9.0) | 65.0 (10.8) | 59.0 (14.3) | 64.1 (13.6) | 66.5 (3.5) | 64.2 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 5 | 0 | 9 | 1 | 29
  Male | 35 | 22 | 16 | 6 | 8 | 1 | 88

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Adverse Events (AEs) Who Underwent Percutaneous Coronary Interventions (PCI)
Description: An AE is any unfavorable and unintended change in the structure, function or chemistry of the body temporally associated with study drug administration, whether or not considered related to the study drug.
Time Frame: Up to Day 60
Population: The population included all enrolled participants who received at least 1 dose of study drug and underwent PCI.
Measure: Number; unit: Participants
Groups:
- Vorapaxar 20 mg Loading Dose PCI: Vorapaxar 20 mg as a loading dose is administered as the initial dose. From Day 2, 1mg or 2.5 mg once daily is administered as the maintenance dose for 59 days (total duration of 60 days).
- Vorapaxar 40 mg Loading Dose PCI: Vorapaxar 40 mg as a loading dose is administered as the initial dose. From Day 2, 1 mg or 2.5 mg once daily is administered as the maintenance dose for 59 days (total duration of 60 days).
- Placebo/Placebo PCI: Placebo as loading dose is administered as the initial dose. From Day 2, placebo once daily is administered as the maintenance dose for 59 days (total duration of 60 days).
Arm/Group | Vorapaxar 20 mg Loading Dose PCI | Vorapaxar 40 mg Loading Dose PCI | Placebo/Placebo PCI
Number analyzed (Participants) | 40 | 31 | 21
Participants | 40 | 30 | 21

2. Secondary Outcome: Number of Participants Experiencing Non-Major Adverse Cardiac Events (MACE) Who Underwent PCI
Description: An AE is any unfavorable and unintended change in the structure, function or chemistry of the body temporally associated with study drug administration, whether or not considered related to the study drug. MACE events were defined as nonfatal myocardial infarction (MI), nonfatal stroke, hospitalization due to recurrent ischemia, or urgent coronary revascularization performed ≥ 30 days after administration of the loading dose (Day 1). All MACE events were excluded from this analysis. Analysis of data was by loading/maintenance dose group.
Time Frame: Up to Day 121
Population: The population included all enrolled participants who received at least 1 dose of study drug and underwent PCI with Non-Major MACE data available.
Measure: Number; unit: Participants
Groups:
- Vorapaxar 20 mg/1 mg PCI: Vorapaxar 20 mg as loading dose is administered as the initial dose. From Day 2, 1 mg once daily is administered as the maintenance dose for 59 days (total duration of 60 days).
- Vorapaxar 20 mg/2.5 mg PCI: Vorapaxar 20 mg as loading dose is administered as the initial dose. From Day 2, 2.5 mg once daily is administered as the maintenance dose for 59 days (total duration of 60 days).
- Vorapaxar 40 mg/1 mg PCI: Vorapaxar 40 mg as loading dose is administered as the initial dose. From Day 2, 1 mg once daily is administered as the maintenance dose for 59 days (total duration of 60 days).
- Vorapaxar 40 mg/2.5 mg PCI: Vorapaxar 40 mg as loading dose is administered as the initial dose. From Day 2, 2.5 mg once daily is administered as the maintenance dose for 59 days (total duration of 60 days).
Arm/Group | Vorapaxar 20 mg/1 mg PCI | Vorapaxar 20 mg/2.5 mg PCI | Vorapaxar 40 mg/1 mg PCI | Vorapaxar 40 mg/2.5 mg PCI | Placebo/Placebo PCI
Number analyzed (Participants) | 21 | 19 | 16 | 15 | 21
Participants | 21 | 19 | 16 | 14 | 21

3. Secondary Outcome: Number of Participants With Major, Minor, and Non-Thrombolysis in Myocardial Infarction Cooperative Group (TIMI) Bleeding Events Among Participants Who Underwent PCI
Description: Major TIMI bleeding was defined as any intracranial bleeding (excluding microhemorrhages <10 mm evident only on gradient-echo magnetic resonance imaging [MRI]), clinically overt signs of hemorrhage associated with a drop in hemoglobin of ≥5 g/dL, or fatal bleeding (bleeding that directly results in death within 7 days). Minor TIMI bleeding was defined as any clinically overt bleeding resulting in hemoglobin drop of 3 to <5 g/dL. Non-TIMI bleeding included all bleeding events not covered under Major TIMI bleeding or Minor TIMI bleeding. Analysis of data was by maintenance dose group.
Time Frame: Up to Day 60
Population: The population included all enrolled participants who received at least 1 dose of study drug and underwent PCI with TIMI bleeding data available.
Measure: Number; unit: Participants
Groups:
- Vorapaxar 1 mg Maintenance Dose PCI: Vorapaxar 20 mg or 40 mg as loading dose is administered as the initial dose. From Day 2, 1 mg once daily is administered as the maintenance dose for 59 days (total duration of 60 days).
- Vorapaxar 2.5 mg Maintenance Dose PCI: Vorapaxar 20 mg or 40 mg as loading dose is administered as the initial dose. From Day 2, 1 mg or 2.5 mg once daily is administered as the maintenance dose for 59 days (total duration of 60 days).
Arm/Group | Vorapaxar 1 mg Maintenance Dose PCI | Vorapaxar 2.5 mg Maintenance Dose PCI | Placebo/Placebo PCI
Number analyzed (Participants) | 37 | 33 | 21
Participants
  Major TIMI Bleeding Events | 2 | 0 | 0
  Minor TIMI Bleeding Events | 5 | 3 | 2
  Non-TIMI Bleeding Events | 22 | 17 | 11

4. Secondary Outcome: Number of Participants Who Underwent PCI With Inhibition of Platelet Aggregation By Study Visit
Description: Blood samples were collected from participants at Baseline and Days 30, 60, 74, 90, and 121 to determine the extent of inhibition of platelet aggregation induced by thrombin-receptor agonist peptide (TRAP). Analysis of data was by maintenance dose group.
Time Frame: Baseline, Day 30, Day 60, Day 74, Day 90, Day 121
Population: The population consisted of all enrolled participants who received at least 1 dose of study drug and underwent PCI with inhibition of platelet aggregation data available.
Measure: Number; unit: Participants
Groups:
- Vorapaxar 2.5 mg Maintenance Dose PCI: Vorapaxar 20 mg or 40 mg as loading dose is administered as the initial dose. From Day 2, 2.5 mg once daily is administered as the maintenance dose for 59 days (total duration of 60 days).
Arm/Group | Vorapaxar 1 mg Maintenance Dose PCI | Vorapaxar 2.5 mg Maintenance Dose PCI | Placebo/Placebo PCI
Number analyzed (Participants) | 5 | 4 | 3
Participants
  Baseline | 5 | 4 | 3
  Day 30 | 5 | 4 | 3
  Day 60 | 3 | 3 | 1
  Day 74 (follow-up period) | 5 | 4 | 3
  Day 90 (follow-up period) | 5 | 4 | 3
  Day 121 (follow-up period) | 5 | 4 | 3

5. Secondary Outcome: Median High-Sensitivity C-Reactive Protein (Hs-CRP) Levels Among Participants Who Underwent PCI By Study Visit
Description: Participant blood samples were collected at Baseline and on Days 30 and 60 to evaluate the median level of hs-CRP. hs-CRP is a protein marker in the blood associated with inflammation with higher values indicating a greater degree of inflammation. Analysis of data was by maintenance dose group.
Time Frame: Baseline, Day 30, Day 60
Population: The population included all enrolled participants who received at least 1 dose of study drug and underwent PCI with hs-CRP data available.
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Vorapaxar 1 mg Maintenance Dose PCI | Vorapaxar 2.5 mg Maintenance Dose PCI | Placebo/Placebo PCI
Number analyzed (Participants) | 37 | 34 | 21
mg/L
  Baseline (n=37, 34, 21) | 1.30 [0.54 to 4.50] | 2.00 [0.61 to 8.36] | 1.78 [0.66 to 4.50]
  Day 30 (n=35, 34, 21) | 1.28 [0.43 to 7.90] | 1.01 [0.70 to 5.62] | 2.99 [1.14 to 9.40]
  Day 60 (n=30, 25, 13) | 1.20 [0.39 to 3.00] | 0.79 [0.44 to 2.02] | 1.27 [0.61 to 4.88]

6. Secondary Outcome: Mean CD40 Ligand Levels Among Participants Who Underwent PCI
Description: Participant blood samples were collected at Baseline and Days 30 and 60 to evaluate the mean level of CD40 ligand present. CD40 ligand is a protein primarily found on activated T-cells, with higher levels indicating better immunological health. Analysis of data was by maintenance dose group.
Time Frame: Baseline, Day 30, Day 60
Population: The population included all enrolled participants who received at least 1 dose of study drug and underwent PCI with CD40 ligand data available.
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Vorapaxar 1 mg Maintenance Dose PCI | Vorapaxar 2.5 mg Maintenance Dose PCI | Placebo/Placebo PCI
Number analyzed (Participants) | 37 | 34 | 21
ng/mL
  Baseline (n=37, 34, 21) | 5.6 (0.56) [0.54 to 4.50] | 6.9 (0.60) [0.61 to 8.36] | 4.8 (0.79) [0.66 to 4.50]
  Day 30 (n=35, 34, 31) | 5.9 (0.52) [0.43 to 7.90] | 5.9 (0.63) [0.70 to 5.62] | 6.2 (0.73) [1.14 to 9.40]
  Day 60 (n=30, 25, 13) | 5.6 (0.55) [0.39 to 3.00] | 5.4 (0.58) [0.44 to 2.02] | 5.7 (1.21) [0.61 to 4.88]

7. Secondary Outcome: Mean Membrane-Bound P-Selectin Levels Among Participants Who Underwent PCI
Description: Participant blood samples were collected at Baseline and Days 30 and 60 to evaluate the mean level of membrane-bound P-selectin. Membrane-bound P-selectin was measured using flow cytometry and a monoclonal antibody to P-selectin. Intensity levels are reported in arbitrary units 0 (dark) to 1023 (bright). Higher values correspond to greater membrane-bound P-Selectin levels. Analysis of data was by maintenance dose group.
Time Frame: Baseline, Day 30, Day 60
Population: The population included all enrolled participants that received at least 1 dose of study drug and underwent PCI with membrane-bound P-selectin data available.
Measure: Mean (Standard Error); unit: Arbitrary Units
Arm/Group | Vorapaxar 1 mg Maintenance Dose PCI | Vorapaxar 2.5 mg Maintenance Dose PCI | Placebo/Placebo PCI
Number analyzed (Participants) | 4 | 4 | 3
Arbitrary Units
  Baseline (n=4, 4, 3) | 24.8 (2.86) [0.54 to 4.50] | 16.5 (0.83) [0.61 to 8.36] | 15.9 (1.25) [0.66 to 4.50]
  Day 30 (n=3, 4, 3) | 20.6 (1.76) [0.43 to 7.90] | 16.4 (0.85) [0.70 to 5.62] | 18.8 (0.91) [1.14 to 9.40]
  Day 60 (n=2, 3, 1) | 25.0 (2.80) [0.39 to 3.00] | 14.9 (0.62) [0.44 to 2.02] | 19.4 (NA) [0.61 to 4.88] — SE not calculable since n=1.

8. Secondary Outcome: Number of Participants Who Underwent PCI With Clinically Important Bleeding Events During Treatment and After Hospital Discharge
Description: Clinically important bleeding events were defined as intracranial hemorrhage, bleeding requiring hospitalization, or TIMI major bleeding. Analysis of data was by loading/maintenance dose group.
Time Frame: Up to Day 121
Population: The population included all participants who received at least 1 dose of study drug, underwent PCI, and had bleeding event data.
Measure: Number; unit: Participants
Arm/Group | Vorapaxar 20 mg/1 mg PCI | Vorapaxar 20 mg/2.5 mg PCI | Vorapaxar 40 mg/1 mg PCI | Vorapaxar 40 mg/2.5 mg PCI | Placebo/Placebo PCI
Number analyzed (Participants) | 21 | 19 | 16 | 15 | 21
Participants
  Treatment Phase | 3 | 0 | 2 | 0 | 0
  Post-Hospital Discharge | 1 | 0 | 2 | 0 | 0

9. Secondary Outcome: Number of Participants With Major, Minor, and Non-TIMI Bleeding Events Among Participants Who Did Not Undergo PCI
Description: Major TIMI bleeding was defined as any intracranial bleeding (excluding microhemorrhages <10 mm evident only on gradient-echo MRI), clinically overt signs of hemorrhage associated with a drop in hemoglobin of ≥5 g/dL, or fatal bleeding (bleeding that directly results in death within 7 days). Minor TIMI bleeding was defined as any clinically overt bleeding resulting in hemoglobin drop of 3 to <5 g/dL. Non-TIMI bleeding included all bleeding events not covered under Major TIMI bleeding or Minor TIMI bleeding. Analysis of data was by loading dose group.
Time Frame: Up to Day 60
Population: The population consisted of all enrolled participants who received at least 1 dose of study drug, did not undergo PCI, and had TIMI bleeding data available.
Measure: Number; unit: Participants
Groups:
- Vorapaxar 20 mg Loading Dose Non-PCI: Vorapaxar 20 mg as a loading dose is administered as the initial dose. From Day 2, 1mg or 2.5 mg once daily is administered as the maintenance dose for 59 days (total duration of 60 days).
- Vorapaxar 40 mg Loading Dose Non-PCI: Vorapaxar 40 mg as a loading dose is administered as the initial dose. From Day 2, 1 mg or 2.5 mg once daily is administered as the maintenance dose for 59 days (total duration of 60 days).
- Placebo/Placebo Non-PCI: Placebo as loading dose is administered as the initial dose. From Day 2, placebo once daily is administered as the maintenance dose for 59 days (total duration of 60 days).
Arm/Group | Vorapaxar 20 mg Loading Dose Non-PCI | Vorapaxar 40 mg Loading Dose Non-PCI | Placebo/Placebo Non-PCI
Number analyzed (Participants) | 6 | 17 | 2
Participants
  Major TIMI Events | 1 | 2 | 0
  Minor TIMI Events | 0 | 0 | 0
  Non-TIMI Bleeding Events | 1 | 8 | 1

10. Secondary Outcome: Number of Participants Experiencing Non-MACE AEs Among Participants Who Did Not Undergo PCI
Description: An AE is any unfavorable and unintended change in the structure, function or chemistry of the body temporally associated with study drug administration, whether or not considered related to the study drug. MACE events were defined as nonfatal MI, nonfatal stroke, hospitalization due to recurrent ischemia, or urgent coronary revascularization performed ≥ 30 days after administration of the loading dose (Day 1). All MACE events were excluded from this analysis. Analysis of data was by loading dose group.
Time Frame: Up to Day 121
Population: The population consisted of all enrolled participants who received at least 1 dose of study drug, did not undergo PCI, and had non-MACE AE data available.
Measure: Number; unit: Participants
Arm/Group | Vorapaxar 20 mg Loading Dose Non-PCI | Vorapaxar 40 mg Loading Dose Non-PCI | Placebo/Placebo Non-PCI
Number analyzed (Participants) | 6 | 17 | 2
Participants | 6 | 15 | 1

11. Secondary Outcome: Number of Participants Who Did Not Undergo PCI But Had Coronary Artery Bypass Graft (CABG) Who Experienced Bleeding Events
Description: Bleeding events were evaluated up to 10 hours post-CABG among participants who did not undergo PCI.
Time Frame: Up to 10 Hours Post-CABG
Population: Evaluation of the bleeding events associated with CABG occurring after Vorapaxar treatment was not analyzed since only three participants in the non-PCI cohort underwent CABG in this study.
Arm/Group | Vorapaxar 20 mg Loading Dose Non-PCI | Vorapaxar 40 mg Loading Dose Non-PCI | Placebo/Placebo Non-PCI
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Number of Participants Who Did Not Undergo PCI But Had Bleeding Events That Required Transfusion
Description: Bleeding events were evaluated among participants that did not undergo PCI to determine the number of participants that required blood transfusion. Analysis of data was by loading dose group.
Time Frame: Up to Day 60
Population: The population consisted of all enrolled participants who received at least 1 dose of study drug, did not undergo PCI, and had transfusion data available.
Measure: Number; unit: Participants
Arm/Group | Vorapaxar 20 mg Loading Dose Non-PCI | Vorapaxar 40 mg Loading Dose Non-PCI | Placebo/Placebo Non-PCI
Number analyzed (Participants) | 6 | 17 | 2
Participants | 1 | 2 | 0

13. Secondary Outcome: Number of Participants Who Did Not Undergo PCI But Had Bleeding Events That Required Subsequent Hospitalization
Description: Bleeding events were evaluated among participants that did not undergo PCI to determine the number of participants who required a subsequent hospitalization. Analysis of data was by loading dose group.
Time Frame: Up to Day 30
Population: The population consisted of all enrolled participants who received at least 1 dose of study drug, did not undergo PCI, and had hospitalization data available.
Measure: Number; unit: Participants
Arm/Group | Vorapaxar 20 mg Loading Dose Non-PCI | Vorapaxar 40 mg Loading Dose Non-PCI | Placebo/Placebo Non-PCI
Number analyzed (Participants) | 6 | 17 | 2
Participants | 0 | 1 | 0

14. Secondary Outcome: Median Hs-CRP Levels Among Participants Who Did Not Undergo PCI
Description: Participant blood samples were collected at baseline and at the time of hospital discharge to determine the median serum level of hs-CRP. Analysis of data was by loading dose group.
Time Frame: Baseline Up To Day 60
Population: The population consisted of all enrolled participants who received at least 1 dose of study drug, did not undergo PCI, and had hs-CRP data available.
Measure: Median (Standard Deviation); unit: mg/L
Arm/Group | Vorapaxar 20 mg Loading Dose Non-PCI | Vorapaxar 40 mg Loading Dose Non-PCI | Placebo/Placebo Non-PCI
Number analyzed (Participants) | 6 | 17 | 2
mg/L
  Baseline | 2.57 (5.70) | 1.05 (2.23) | 6.94 (12.01)
  Time of Hospital Discharge | 3.56 (10.12) | 2.65 (5.00) | 3.96 (0.91)

15. Secondary Outcome: Mean CD40 Ligand Levels Among Participants Who Did Not Undergo PCI
Description: Participant blood samples were collected at baseline and at the time of hospital discharge to determine the mean serum level of CD40 ligand. Analysis of data was by loading dose group.
Time Frame: Baseline Up To Day 60
Population: The population consisted of all enrolled participants who received at least 1 dose of study drug, did not undergo PCI, and had CD40 ligand data available.
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Vorapaxar 20 mg Loading Dose Non-PCI | Vorapaxar 40 mg Loading Dose Non-PCI | Placebo/Placebo Non-PCI
Number analyzed (Participants) | 6 | 17 | 2
ng/mL
  Baseline | 8.4 (1.10) | 4.6 (0.79) | 11.1 (4.06)
  Time of Hospital Discharge | 10.1 (2.86) | 7.1 (0.83) | 12.9 (4.64)

16. Secondary Outcome: Number of Participants Who Did Not Undergo PCI That Had Clinically Important Bleeding Events
Description: Clinically important bleeding events were defined as intracranial hemorrhage, bleeding requiring blood transfusion, bleeding requiring hospitalization, and TIMI major bleeding. Analysis of data was by loading dose group.
Time Frame: Baseline Up To Day 60
Population: The population consisted of all enrolled participants who received at least 1 dose of study drug, did not undergo PCI, and had bleeding event data available.
Measure: Number; unit: Participants
Arm/Group | Vorapaxar 20 mg Loading Dose Non-PCI | Vorapaxar 40 mg Loading Dose Non-PCI | Placebo/Placebo Non-PCI
Number analyzed (Participants) | 6 | 17 | 2
Participants
  Intracranial hemorrhage | 0 (1.10) | 1 (0.79) | 0 (4.06)
  Bleeding requiring transfusion | 1 (2.86) | 2 (0.83) | 0 (4.64)
  Bleeding requiring hospitalization | 0 | 1 | 0
  Major TIMI bleeding | 1 | 2 | 0

ADVERSE EVENTS:
Time Frame: Up to Day 121
Description: As this was a safety study of Vorapaxar in a clinical setting administered concomitantly with other antiplatelet agents, safety data were collected for all 120 enrolled participants on study, regardless of treatment with study drug.
Groups:
- Vorapaxar 20 mg/1 mg: Vorapaxar 20 mg as loading dose is administered as the initial dose. From Day 2, 1 mg once daily is administered as the maintenance dose for 59 days (total duration of 60 days).
- Vorapaxar 20 mg/2.5 mg: Vorapaxar 20 mg as loading dose is administered as the initial dose. From Day 2, 2.5 mg once daily is administered as the maintenance dose for 59 days (total duration of 60 days).
- Vorapaxar 40 mg/1 mg: Vorapaxar 40 mg as loading dose is administered as the initial dose. From Day 2, 1 mg once daily is administered as the maintenance dose for 59 days (total duration of 60 days).
- Vorapaxar 40 mg/2.5 mg: Vorapaxar 40 mg as loading dose is administered as the initial dose. From Day 2, 2.5 mg once daily is administered as the maintenance dose for 59 days (total duration of 60 days).
- Placebo/Placebo: Placebo as loading dose is administered as the initial dose. From Day 2, placebo once daily is administered as the maintenance dose for 59 days (total duration of 60 days).
Arm/Group | Vorapaxar 20 mg/1 mg | Vorapaxar 20 mg/2.5 mg | Vorapaxar 40 mg/1 mg | Vorapaxar 40 mg/2.5 mg | Placebo/Placebo
Serious Adverse Events (participants affected / at risk) | 5/25 | 4/24 | 2/22 | 2/26 | 5/23
Other Adverse Events (participants affected / at risk) | 25/25 | 23/24 | 22/22 | 23/26 | 22/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorapaxar 20 mg/1 mg (N=25) | Vorapaxar 20 mg/2.5 mg (N=24) | Vorapaxar 40 mg/1 mg (N=22) | Vorapaxar 40 mg/2.5 mg (N=26) | Placebo/Placebo (N=23)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac Tamponade (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricle Rupture (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sudden Hearing Loss (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaena (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest Discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood Glucose Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colon Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Loss of Consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subarachnoid Haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal Failure Acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arteriosclerosis Obliterans (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorapaxar 20 mg/1 mg (N=25) | Vorapaxar 20 mg/2.5 mg (N=24) | Vorapaxar 40 mg/1 mg (N=22) | Vorapaxar 40 mg/2.5 mg (N=26) | Placebo/Placebo (N=23)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (2) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 3 (3) | 3 (3) | 5 (5) | 2 (2) | 9 (10)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Ventricular Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Abdominal Distention (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 6 (7) | 7 (8) | 3 (3) | 4 (5) | 6 (7)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Gingival Bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Periodontitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 1 (1)
Chest Discomfort (General disorders) | 3 (3) | 3 (3) | 3 (4) | 4 (4) | 2 (2)
Chest Pain (General disorders) | 2 (2) | 3 (9) | 1 (1) | 2 (2) | 2 (2)
Oedema Peripheral (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Puncture Site Haemorrhage (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Puncture Site Pain (General disorders) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 6 (7) | 3 (3) | 3 (3) | 0 (0) | 3 (3)
Venipuncture Site Swelling (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic Function Abnormal (Hepatobiliary disorders) | 2 (2) | 1 (1) | 2 (2) | 5 (5) | 3 (3)
Gingival Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 4 (5) | 4 (4) | 5 (5) | 2 (3) | 3 (3)
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 2 (2) | 2 (3) | 4 (5)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 3 (3) | 3 (3) | 4 (4)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood Alkaline Phosphatase Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Blood Creatine Phosphokinase Increased (Investigations) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Blood Creatinine Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blood Pressure Decreased (Investigations) | 2 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Pressure Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Blood Triglycerides Increased (Investigations) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 0 (0)
Blood Urine Present (Investigations) | 4 (5) | 1 (1) | 2 (3) | 3 (3) | 2 (3)
Gamma-Glutamyltransferase Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 2 (2)
Haemoglobin Decreased (Investigations) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 2 (3)
Occult Blood (Investigations) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Occult Blood Positive (Investigations) | 12 (13) | 8 (8) | 10 (10) | 7 (9) | 10 (10)
Protein Urine Present (Investigations) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
White Blood Cell Count Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Hyperchlesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 7 (8) | 3 (3) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 1 (3) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Dizziness Postural (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 5 (5) | 3 (3) | 5 (5)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 5 (5) | 3 (3) | 2 (2) | 7 (7) | 3 (3)
Restlessness (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Oliguria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 4 (5) | 0 (0) | 4 (4) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Cold Sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Drug Eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage Subcutaneous (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 4 (4) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Rash Erythematous (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Angiopathy (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 2 (2) | 5 (6) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior approval by the Sponsor is required before the results obtained in the clinical study can be made public by the investigator (sub-investigator) in a publication or at a medical meeting.